CLINICAL TRIAL: NCT02991443
Title: The Effect of Mindfulness Based Stress Reduction on Parents of Children With Inflammatory Bowel Disease
Brief Title: Mindfulness Based Stress Reduction for Parents of Children With IBD
Acronym: Mindful
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MindfulnessSMCIBD
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness based stress reduction (Experimental): Parents of children with IBD will undergo mindfulness based stress reduction (MBSR) intervention consisted of 8 group sessions. The effect on stress and anxiety will be assessed using 3 validated questionnaires which will be filled prior to intervention, at the end of intervention and 3 months following intervention.
  Interventions: Behavioral: Mindfulness based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — Mindfulness based stress reduction consisted of 8 group sessions for parents of children with IBD

SUMMARY:
Parents of children with chronic diseases often report increased level of stress and anxiety. The aim of the study is to assess the effect of mindfulness based stress reduction (MBSR) intervention on stress and anxiety of parents of children with inflammatory bowel diseases (IBD). The intervention is consisted of 8 group sessions managed by a certified psychologist. 30 parents will participate. The efficacy of the intervention will be assessed by 3 validated questionnaires which will be filled by each participant prior to intervention, at the end of intervention and 3 months following interventions.

DETAILED DESCRIPTION:
Parents of children with chronic diseases often report increased level of stress and anxiety. Inflammatory bowel diseases (IBD), including crohn's disease and ulcerative colitis are chronic debilitating conditions with significant implications of both patients and parents. Thus, there is a necessity to address the stress and anxiety derived from parenting a child with IBD.

Mindfulness is the psychological process of bringing one's attention to the internal and external experiences occurring in the present moment,which can be developed through the practice of meditation and other training. Clinical studies have documented both physical and mental health benefits of mindfulness in different patient categories as well as in healthy adults and children.

The aim of the study is to assess the effect of mindfulness based stress reduction (MBSR) intervention on stress and anxiety of parents of children with inflammatory bowel diseases (IBD). The intervention is consisted of 8 group sessions managed by a certified psychologist. 30 parents will participate in 4 separated courses. The efficacy of the intervention will be assessed by 3 validated questionnaires which will be filled by each participant prior to intervention, at the end of intervention and 3 months following interventions: Profile of mood states (POMS), The brief symptom inventory (BSI) and perceived stress scale (PSS). Differences in questionnaires' scores will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* A parent to an IBD patient who is younger than 18 years of age

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
The change in perceived stress scale | At baseline and 3 months following intervention

SECONDARY OUTCOMES:
The change in profile of mood states (POMS) score | At week 0 following intervention and 3 months following intervention compared with baseline
The change in brief symptom inventory (BSI) score | At week 0 following intervention and 3 months following intervention compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, MD, Study Director — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No